CLINICAL TRIAL: NCT01157481
Title: Diastolic Heart Failure Management by Nifedipine
Acronym: DEMAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Demand Investigators (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEMAND-01; UMIN000003856 (Other: University hospital Medical Information Network)
Record Dates: First submitted 2010-07-01; First posted 2010-07-07 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Diastolic Heart Failure
Keywords: Diastolic Heart Failure; Heart failure with preserved ejection fraction; nifedipine
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional therapy plus nifedipine (Experimental)
  Interventions: Drug: Conventional therapy plus nifedipine
- Conventional therapy (Active Comparator)
  Interventions: Drug: Conventional therapy

INTERVENTIONS:
Drug: Conventional therapy plus nifedipine — Participants will receive 10 to 60 mg of sustained-release nifedipine once a day until December 2014
  Arms: Conventional therapy plus nifedipine
Drug: Conventional therapy — Conventional therapy
  Arms: Conventional therapy

SUMMARY:
Patients with heart failure with preserved ejection fraction have a equally high risk for mortality and re-hospitalization as those with reduced ejection fraction. Effective management strategies are critically needed to be established for this type of heart failure. These patients have more hypertensive and ischemic etiology than those with reduced ejection fraction. The investigators hypothesis is that Ca channel blocker nifedipine can improve the heart failure clinical composite response endpoint compared with the conventional treatment in patients with heart failure with hypertension and/or coronary artery disease and preserved ejection fraction (>=50%) by echocardiography. This study is multi-center, prospective, randomized, open-label, and blinded-endpoint design.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years and older
2. Heart failure with history of hypertension and/or coronary artery disease
3. LVEF > or = 50% on echocardiography

Exclusion Criteria:

1. Valvular heart diseases with significant regurgitation and/or stenosis
2. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, and active myocarditis
3. Constrictive pericarditis
4. Cardiogenic shock
5. Planned coronary artery bypass grafting or percutaneous coronary intervention within 3 months
6. History of acute coronary syndrome or stroke within 3 months
7. Pregnancy or breastfeeding
8. Hypersensitivity or contraindication to nifedipine
9. Inability to obtain informed consent
10. Any conditions not suitable for the participation in this trial judged by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2010-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Heart failure clinical composite response endpoint | up to 53 months

SECONDARY OUTCOMES:
Death | up to 53 months
Cardiovascular death | up to 53 months
Hospital admission | up to 53 months
Hospital admission for cardiovascular disease | up to 53 months
Hospital admission for worsening heart failure | up to 53 months
Hospital admission for acute myocardial infarction, angina, coronary artery bypass grafting and percutaneous coronary intervention | up to 53 months
Stroke | up to 53 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hokkaido Univestity Hospital, Sapporo, Japan